CLINICAL TRIAL: NCT00995371
Title: Comparative Study of Epidural Steroid Injection Versus Mild® (Minimally Invasive Lumbar Decompression) Procedure in Patients Diagnosed With Symptomatic Moderate to Severe Lumbar Central Canal Stenosis
Brief Title: Study of Epidural Steroid Injection (ESI) Versus Minimally Invasive Lumbar Decompression (Mild®) in Patients With Symptomatic Lumbar Central Canal Stenosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coastal Orthopedics & Sports Medicine (Other)
Collaborators: Vertos Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VMD001LB
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Results first posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-09

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Spinal Stenosis; Lumbar Spinal Stenosis; Laminotomy; Laminectomy; Spine Surgery
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vertos mild® Minimally-Invasive Lumbar Decompression (Active Comparator): Patients in the Vertos mild® treatment group will be treated by appropriately trained physicians in accordance with the product labeling and indications for use.
  Interventions: Device: MILD® (Minimally Invasive Lumbar Decompression)
- Epidural Steroid Injection (Active Comparator): Patients in the Epidural Steroid Injection (ESI) group will have ESI performed by appropriately trained physicians in accordance with product labeling and indications for use.
  Interventions: Drug: Epidural Steroid Injection

INTERVENTIONS:
Device: MILD® (Minimally Invasive Lumbar Decompression) — Image guided minimally-invasive lumbar decompression performed with arthroscopic devices.
  Arms: Vertos mild® Minimally-Invasive Lumbar Decompression
Drug: Epidural Steroid Injection — An Epidural Steroid Injection is injected into the space around the spinal cord and nerve roots called epidural space.
  Arms: Epidural Steroid Injection

SUMMARY:
This is a single-center, randomized, prospective, double-blind clinical study to assess the clinical application and outcomes with MILD® devices versus epidural steroid injection in patients with symptomatic moderate to severe central canal spinal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Lumbar Spinal Stenosis (LSS) primarily caused by dorsal element hypertrophy.
* Prior failure of conservative therapy and ODI Score >20%.
* Radiologic evidence of LSS (L3-L5), Ligamentum flavum >2.5mm, confirmed by pre-op MRI and/or CT.
* Central canal cross sectional area ≤ 100 square mm.
* Anterior listhesis ≤ 5.0mm.
* Able to walk at least 10 feet unaided before being limited by pain.
* Available to complete 26 weeks of follow-up.
* A signed Informed Consent Form is obtained from the patient.
* Adults at least 18 years of age.

Exclusion Criteria:

* Prior surgery at intended treatment level.
* History of recent spinal fractures with concurrent pain symptoms.
* Disabling back or leg pain from causes other than LSS (e.g. acute compression fracture, metabolic neuropathy, or vascular claudication symptoms, etc.)
* Significant / symptomatic disc protrusion or osteophyte formation.
* Excessive / symptomatic facet hypertrophy.
* Bleeding disorders and/or current use of anti-coagulants.
* Use of ASA and/or NSAID within 5 days of treatment.
* Pregnant and/or breastfeeding.
* Epidural steroids previously administered (not ESI naive)
* Wound healing pathologies deemed to compromise outcomes, including: diabetes, excessive smoking history, cancer, connective tissue diseases, recent spine radiation and severe COPD.
* Dementia and/or inability to give informed consent.
* Inability of the patient to lie prone for any reason with anesthesia support (e.g. COPD, obesity, etc.).
* On Workman's Compensation or considering litigation associated with back pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-08; Primary Completion 2012-06 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lora Brown, MD, Principal Investigator — Coastal Orthopedics & Sports Medicine
Locations (1):
- Coastal Orthopedics & Sports Medicine, Bradenton, Florida, United States

REFERENCES:
- [Derived] Brown LL. A double-blind, randomized, prospective study of epidural steroid injection vs. the mild(R) procedure in patients with symptomatic lumbar spinal stenosis. Pain Pract. 2012 Jun;12(5):333-41. doi: 10.1111/j.1533-2500.2011.00518.x. Epub 2012 Jan 25. PMID 22272730

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled through one site (Coastal Orthopedics) between September 2009 and January 2011.
Pre-assignment Details: Randomization occurred in blocks of four. After Week 6 post-treatment and prior to 4 months, ESI arm participants were allowed to cross over to mild if they chose to have it.
Groups:
- Vertos Mild® Minimally-Invasive Lumbar Decompression (Mild): Group 1: Patients in the Vertos mild treatment group will be treated by appropriately trained physicians in accordance with the product labeling and indications for use.
- Epidural Steroid Injection Then Lumbar Decompression With Mild: Group 2: After post-treatment Week 6 and prior to 4 months patients in ESI procedure arm, when unblinded, were given option to cross-over to and receive the mild procedure using the mild device kit
Period: Prior to ESI Cross-over, 6 Weeks
Arm/Group | Vertos Mild® Minimally-Invasive Lumbar Decompression (Mild) | Epidural Steroid Injection Then Lumbar Decompression With Mild
Started | 21 | 17
Completed | 21 | 17
Not Completed | 0 | 0
Period: After ESI Cross-over to Mild, 26 Weeks
Arm/Group | Vertos Mild® Minimally-Invasive Lumbar Decompression (Mild) | Epidural Steroid Injection Then Lumbar Decompression With Mild
Started | 21 | 17
Completed | 16 (All 21 completed Wk 6 Intent to Treat analysis. Sixteen reported Week 26 outcomes.) | 12 (All 17 completed Wk 6 Intent to Treat analysis prior to x-over. After x-over 12 reported Wk 26)
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 5 | 5

BASELINE CHARACTERISTICS:
Population: ITT analysis includes all patients at weeks 6 post-treatment. Week 26 cohort analysis includes 16 mild patients who reported outcomes at Week 26 and the 12 ESI patients who reported outcomes at Week 26 after cross-over to mild.
Groups:
- Epidural Steroid Injection: Group 2: Patients in the Epidural Steroid Injection (ESI) group will be treated by the physicians in accordance with product labeling and indications for use.
- Total: Total of all reporting groups
Arm/Group | Vertos Mild® Minimally-Invasive Lumbar Decompression (Mild) | Epidural Steroid Injection | Total
Number analyzed (Participants) | 21 | 17 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 1 | 6
  >=65 years | 16 | 16 | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 74.24 (10.12) | 78.71 (7.11) | 76.26 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 13 | 8 | 21
Region of Enrollment [Number; unit: participants]
  United States | 21 | 17 | 38

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in VAS
Description: Visual Analog Scale (VAS) - a validated ten point scale where ten is the worst possible pain and zero represents complete lack of pain. The change from baseline to 6 weeks for all participants is presented below, where a positive value represents the baseline value minus the 6 week value.
Time Frame: Baseline and 6 weeks prior to cross-over
Population: All 38 participants (21 in mild and 17 in ESI arm) reported VAS at Week 6 post-treatment. All measurements for the ESI group occurred prior to cross-over to the mild procedure. This is Intent to Treat (ITT) analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Epidural Steroid Injection Prior to Cross-Over: Group 2: Patients in the Epidural Steroid Injection (ESI) group will be treated by the physicians in accordance with product labeling and indications for use.
Arm/Group | Vertos Mild® Minimally-Invasive Lumbar Decompression (Mild) | Epidural Steroid Injection Prior to Cross-Over
Number analyzed (Participants) | 21 | 17
units on a scale | 2.52 [1.09 to 3.96] | 0.06 [-1.43 to 1.55]
Statistical Analysis 1: Comparison: Vertos Mild® Minimally-Invasive Lumbar Decompression (Mild); The mean change from baseline was assessed for VAS using a paired t-test. The resulting p-values are to be considered as descriptive statistics. Two-sided test with 5% Type I error was used; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 2.52, 95% CI 2-sided [1.09 to 3.96]
Statistical Analysis 2: Comparison: Epidural Steroid Injection Prior to Cross-Over; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-1.43 to 1.55]

2. Primary Outcome: Mean Change in ODI
Description: Oswestry Disability Index (ODI) measures permanent functional disability using questions regarding activities of daily living (ADL), specifically disturbance in ADL related to chronic back pain. Higher score indicate a 'more limited' life.
  The ten topics of the ODI are rated from zero (no pain/limitation) to five (high pain/very limited physically). Calculated values range from zero (0% disability) to 100 (100% disability). The change from baseline to 6 weeks for all participants is presented below, where a positive value represents the baseline value minus the 6 week value
Time Frame: Baseline and 6 weeks prior to cross-over
Population: All 38 participants (21 in mild and 17 in ESI arm) reported ODI at Week 6 post-treatment. All measurements for the ESI group occurred prior to cross-over to the mild procedure. This is Intent to Treat (ITT) analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Vertos Mild® Minimally-Invasive Lumbar Decompression (Mild) | Epidural Steroid Injection Prior to Cross-Over
Number analyzed (Participants) | 21 | 17
units on a scale | 11.33 [3.35 to 19.31] | 5.65 [-4.12 to 15.41]
Statistical Analysis 1: Comparison: Vertos Mild® Minimally-Invasive Lumbar Decompression (Mild); The mean change from baseline was assessed for ODI using a paired t-test. The resulting p-values are to be considered as descriptive statistics. Two-sided test with 5% Type I error was used; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 11.33, 95% CI 2-sided [3.35 to 19.31]
Statistical Analysis 2: Comparison: Epidural Steroid Injection Prior to Cross-Over; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 5.65, 95% CI [-4.12 to 15.41]

3. Primary Outcome: Mean Change in VAS
Description: Visual Analog Scale (VAS) - a validated ten point scale where ten is the worst possible pain and zero represents complete lack of pain. The change from baseline to 26 weeks for all participants is presented below, where a positive value represents the baseline value minus the 26 week value.
Time Frame: Baseline and 26 weeks After ESI to mild cross-over
Population: Participants who reported Week 26 outcomes. All findings reported below for the ESI group are after cross-over to mild.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Epidural Steroid Injection Then Lumbar Decompression With Mild: Group 2: After post-treatment Week 6 and prior to 4 months patients in ESI procedure arm, after unblinding, were given option to cross-over to and receive the mild procedure using the mild device kit.
Arm/Group | Vertos Mild® Minimally-Invasive Lumbar Decompression (Mild) | Epidural Steroid Injection Then Lumbar Decompression With Mild
Number analyzed (Participants) | 16 | 12
units on a scale | 2.19 [0.61 to 3.77] | 1.00 [-0.66 to 2.66]
Statistical Analysis 1: Comparison: Vertos Mild® Minimally-Invasive Lumbar Decompression (Mild); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 2.19, 95% CI [0.61 to 3.77]
Statistical Analysis 2: Comparison: Epidural Steroid Injection Then Lumbar Decompression With Mild; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 1.00, 95% CI [-0.66 to 2.66]

4. Primary Outcome: Mean Change in ODI
Description: Oswestry Disability Index (ODI) measures permanent functional disability using questions regarding activities of daily living (ADL), specifically disturbance in ADL related to chronic back pain. Higher score indicate a 'more limited' life.
  The ten topics of the ODI are rated from zero (no pain/limitation) to five (high pain/very limited physically). Calculated values range from zero (0% disability) to 100 (100% disability). The change from baseline to 6 weeks for all participants is presented below, where a positive value represents the baseline value minus the 26 week value
Time Frame: Baseline and 26 weeks After ESI to mild cross-over
Population: Participants who reported Week 26 outcomes. All findings reported below for the ESI group are after cross-over to mild.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Vertos Mild® Minimally-Invasive Lumbar Decompression (Mild) | Epidural Steroid Injection Then Lumbar Decompression With Mild
Number analyzed (Participants) | 16 | 12
units on a scale | 16.13 [7.43 to 24.83] | 6.17 [-1.24 to 13.58]
Statistical Analysis 1: Comparison: Vertos Mild® Minimally-Invasive Lumbar Decompression (Mild); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 16.13, 95% CI [7.43 to 24.83]
Statistical Analysis 2: Comparison: Epidural Steroid Injection Then Lumbar Decompression With Mild; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 6.17, 95% CI [-1.24 to 13.58]

ADVERSE EVENTS:
Groups:
- Vertos Mild® Minimally-Invasive Lumbar Decompression: Group 1: Patients in the Vertos mild® treatment group will be treated by appropriately trained physicians in accordance with the product labeling and indications for use.
- Epidural Steroid Injection: Group 2: Patients in the Epidural Steroid Injection (ESI) group will be treated by the physicians in accordance with product labeling and indications for use.
  The ESI group analyzed crossed over to receive the mild procedure after being unblinded. The results are up to 26 weeks post-mild procedure
- ESI Cross-over to Lumbar Decompression With Mild: Group 3: Patients in the Epidural Steroid Injection (ESI) group treated by the physicians in accordance with product labeling and indications for use, crossed over to receive the mild procedure after being unblinded. The results are up to 26 weeks post-mild procedure
Arm/Group | Vertos Mild® Minimally-Invasive Lumbar Decompression | Epidural Steroid Injection | ESI Cross-over to Lumbar Decompression With Mild
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/21 | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No